CLINICAL TRIAL: NCT00666263
Title: A Randomized, Double-Blind, Placebo Controlled, Cross-over Study of the Effectiveness of Immune Globulin Intravenous (Human), 10% (IGIV, 10%) for the Treatment of Multifocal Motor Neuropathy
Brief Title: Study of the Effectiveness of Intravenous Immune Globulin (10%) for the Treatment of Multifocal Motor Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 160604; 2009-013841-27 (EudraCT Number)
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Results first posted 2013-03-13 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Multifocal Motor Neuropathy
MeSH Terms: interventions — gamma-Globulins; Albumins; Solutions; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IGIV, 10% Then Placebo (Experimental): STUDY PART 1: Open-label stabilization on IGIV, 10% (Stabilization Phase 1) all participants. STUDY PART 2: IGIV, 10% (double-blind treatment Cross-Over Period 1). STUDY PART 3: Between the two double-blind treatment cross-over periods, participants received open-label treatment/stabilization with IGIV, 10% (Stabilization Phase 2). STUDY PART 4: Placebo (0.25% human albumin: BUMINATE 25% Albumin (Human)(Baxter Healthcare Corporation) used where licensed; otherwise Human Albumin 200 g/L Baxter Solution for Infusion was used) (double-blind treatment cross-over period 2). STUDY PART 5: Participants received open-label treatment/stabilization with IGIV, 10% (Stabilization Phase 3).
  Each study part was 12 weeks in length. Participants received IGIV, 10% at the same equivalent dose per week administered prior to the study (0.4 to 2.0 g per kg body weight (BW) per infusion cycle).
  Interventions: Biological: Immune Globulin Intravenous (human), 10%; Biological: 0.25% human albumin solution (Placebo)
- Placebo Then IGIV, 10% (Experimental): STUDY PART 1: Open-label stabilization on IGIV, 10% (Stabilization Phase 1) all participants. STUDY PART 2: Placebo (0.25% human albumin: BUMINATE 25% Albumin (Human) (Baxter Healthcare Corporation) used where licensed; otherwise Human Albumin 200 g/L Baxter Solution for Infusion was used) (double-blind treatment Cross-Over Period 1). STUDY PART 3: Between the two double-blind treatment cross-over periods, participants received open-label treatment/stabilization with IGIV, 10% (Stabilization Phase 2). STUDY PART 4: IGIV, 10% (double-blind treatment cross-over period 2). STUDY PART 5: Participants received open-label treatment/stabilization with IGIV, 10% (Stabilization Phase 3).
  Each study part was 12 weeks in length. Participants received IGIV, 10% at the same equivalent dose per week administered prior to the study (0.4 to 2.0 g per kg BW per infusion cycle)
  Interventions: Biological: Immune Globulin Intravenous (human), 10%; Biological: 0.25% human albumin solution (Placebo)

INTERVENTIONS:
Biological: Immune Globulin Intravenous (human), 10% — Dose: Previous dose with 3, 4, or 6 cycles depending on previous schedule (patient specific)
  Other Names: IGIV, 10%; GAMMAGARD LIQUID; KIOVIG
Biological: 0.25% human albumin solution (Placebo) — Cross-over Period 1 (Randomized) / Cross-over Period 2 (opposite of the treatment received in Cross-over Period 1); Dose: Same volume/frequency as Stabilization Phase 1
  Other Names: BUMINATE 25%, Albumin (Human) Solution; Human Albumin 200 g/L Baxter

SUMMARY:
The purpose of the study is to evaluate the efficacy (effect on grip strength and disability) and safety/tolerability of IGIV, 10% in subjects with Multifocal Motor Neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the participant prior to any study-related procedures and study product administration
* Diagnosis of definite or probable MMN based on the criteria of the American Association of Electrodiagnostic Medicine (AAEM) (Olney et al., 2003, see Section 15.1 for the full length publication). Conduction block can be identified by a drop in amplitude. Diagnosis can be based on chart records a) Hand grip (finger flexor) weakness of Medical Research Council (MRC) grade 4 or less at disease onset or appearing prior to screening; b) No upper motor signs c) No bulbar or cranial signs or symptoms; d) No clinically identifiable sensory abnormalities
* Must be on a stable regimen of IGIV for at least 3 months prior to first study product administration
* Treatment interval with IGIV of 2 to 5 weeks (+/- 3 days)
* Dose of IGIV to be 0.4 to 2.0 g per kg BW and infusion cycle
* Participants are adults, male or female, at least 18 years of age
* If female and capable of bearing children - have a negative urine pregnancy test result at enrollment and agree to employ adequate birth control measures for the duration of the study
* Ability and willingness to travel to the study site for infusions and assessments if required by the protocol

Exclusion Criteria:

* Any clinical or electrophysiological evidence of coexisting neuropathy which may interfere with outcome assessments, such as diabetic neuropathy, toxic neuropathy, or neuropathy due to systemic lupus erythematosus
* Treatment with other immunosuppressive agents besides IGIV, which has demonstrated efficacy in MMN such as cyclophosphamide during the 3 months prior to enrollment (or treatment with Rituximab during the 12 months prior to enrollment). Pre-study treatment with mycophenolate mofetil or azathioprine is permitted if the dose has been stable for 3 months prior to enrollment.
* Cerebrospinal fluid protein > 100 mg/dL (if done as part of a previous evaluation)
* Participants positive at enrollment for one or more of the following: Hepatitis B surface antigen (HBsAg), polymerase chain reaction (PCR) for Hepatitis C (HCV), PCR for human immunodeficiency virus (HIV) Type 1
* Participants with levels of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal for the testing laboratory
* Participants with neutropenia (defined as an absolute neutrophil count [ANC]≤1000/mm^3)
* Participants with serum creatinine levels greater than 1.5 times the upper limit of normal for age and gender
* Participants with malignancy other than adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Participants with a history of thrombotic episodes (deep vein thrombosis, myocardial infarction, cerebrovascular accident)
* Participants who received any blood or blood product exposure other than an IGIV, subcutaneous immunoglobulin, immune serum globulin (ISG) preparation, or albumin within the 6 months prior to enrollment
* Participants with an ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following IGIV or human albumin
* Participants with immunoglobulin A (IgA) deficiency and known anti IgA antibodies
* Participants using another investigational product or device within 30 days prior to enrollment
* Participants who are unable or unwilling to meet all the requirements of this study
* If female, is pregnant or lactating at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-08-22 (Actual); Primary Completion 2011-08-11 (Actual); Study Completion 2011-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (17):
- United States (12):
  - Los Angeles, California
  - Stanford, California
  - Centennial, Colorado
  - Miami, Florida
  - Kansas City, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - St Louis, Missouri
  - Columbus, Ohio
  - Portland, Oregon
  - Houston, Texas
  - Seattle, Washington
- Canada (4):
  - Calgary, Alberta
  - Kingston, Ontario
  - London, Ontario
  - Montreal, Quebec
- Aarhus, Denmark

REFERENCES:
- [Background] Merkies IS, Schmitz PI, van der Meche FG, Samijn JP, van Doorn PA; Inflammatory Neuropathy Cause and Treatment (INCAT) group. Clinimetric evaluation of a new overall disability scale in immune mediated polyneuropathies. J Neurol Neurosurg Psychiatry. 2002 May;72(5):596-601. doi: 10.1136/jnnp.72.5.596. PMID 11971045
- [Background] Sharrack B, Hughes RA. The Guy's Neurological Disability Scale (GNDS): a new disability measure for multiple sclerosis. Mult Scler. 1999 Aug;5(4):223-33. doi: 10.1177/135245859900500406. PMID 10467380
- [Result] Koski CL, Schiff RI, Oh M, Lee D. Characteristics of patients with multifocal motor neuropathy enrolled in a randomized controlled trial of intravenous gammaglobulin. Poster. 63rd Annual Meeting of American Academy of Neurology (AAN), April 9-16, 2011, Honolulu, HI, USA.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted in the U.S., Canada, and Europe at 17 study sites. The first participant was enrolled in August 2008.
Pre-assignment Details: Fifty unique potential participants were enrolled at clinical study sites in North America and Europe. Six were screen failures. Therefore, 44 participants were randomized.
Groups:
- IGIV, 10% Then Placebo (During Cross-Over Periods): Each of the following 5 study parts is 12 weeks. Study Part 1: Open-label phase of treatment/stabilization on IGIV, 10% (Stabilization Phase 1) all participants Study Part 2: IGIV, 10% (double-blind treatment cross-over period 1) Study Part 3: Between the two double-blind treatment cross-over periods, participants received open-label treatment/stabilization with IGIV, 10% (Stabilization Phase 2) Study Part 4: Placebo (0.25% human albumin: BUMINATE 25% Albumin (Human)(Baxter Healthcare Corporation) used where licensed; otherwise Human Albumin 200 g/L Baxter Solution for Infusion was used) (double-blind treatment cross-over period 2) Study Part 5: Participants received open-label treatment/stabilization with IGIV, 10% (Stabilization Phase 3)
- Placebo Then IGIV, 10% (During Cross-Over Periods): Each of the following 5 study parts is 12 weeks. Study Part 1: Open-label phase of treatment/stabilization on IGIV, 10% (Stabilization Phase 1) all participants Study Part 2: Placebo (0.25% human albumin: BUMINATE 25% Albumin (Human)(Baxter Healthcare Corporation) used where licensed; otherwise Human Albumin 200 g/L Baxter Solution for Infusion was used) (double-blind treatment cross-over period 1) Study Part 3: Between the two double-blind treatment cross-over periods, participants received open-label treatment/stabilization with IGIV, 10% (Stabilization Phase 2) Study Part 4: IGIV, 10% (double-blind treatment cross-over period 2) Study Part 5: Participants received open-label treatment/stabilization with IGIV, 10% (Stabilization Phase 3)
Period: Study Part 1 (Stabilization Phase 1)
Arm/Group | IGIV, 10% Then Placebo (During Cross-Over Periods) | Placebo Then IGIV, 10% (During Cross-Over Periods)
Started | 22 | 22
Completed | 22 | 21
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Study Part 2 (Cross-over Period 1)
Arm/Group | IGIV, 10% Then Placebo (During Cross-Over Periods) | Placebo Then IGIV, 10% (During Cross-Over Periods)
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0
Period: Study Part 3 (Stabilization Phase 2)
Arm/Group | IGIV, 10% Then Placebo (During Cross-Over Periods) | Placebo Then IGIV, 10% (During Cross-Over Periods)
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0
Period: Study Part 4 (Cross-over Period 2)
Arm/Group | IGIV, 10% Then Placebo (During Cross-Over Periods) | Placebo Then IGIV, 10% (During Cross-Over Periods)
Started | 22 | 21
Completed | 21 | 21
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Study Part 5 (Stabilization Phase 3)
Arm/Group | IGIV, 10% Then Placebo (During Cross-Over Periods) | Placebo Then IGIV, 10% (During Cross-Over Periods)
Started | 21 | 21
Completed | 21 | 20
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: End of Study Visit
Arm/Group | IGIV, 10% Then Placebo (During Cross-Over Periods) | Placebo Then IGIV, 10% (During Cross-Over Periods)
Started | 22 (End of Study Visit done on all 22 randomized regardless of participation in Study Parts) | 22 (End of Study Visit done on all 22 randomized regardless of participation in Study Parts)
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Each participant was to complete 5 study parts (3 stabilization phases of open label treatment with IGIV, 10%, and 1 cross-over period each of double-blind treatment with IGIV, 10% and placebo according to a randomized sequence). Each study part lasted 12 weeks and comprised 3, 4 or 6 infusion cycles depending on treatment interval. Study Part 1: Open-label phase of treatment/stabilization on IGIV, 10% (Stabilization Phase 1) for all participants Study Part 2: Participants were randomized to 1 of 2 sequences of double-blind treatment (either: IGIV, 10% or placebo) Study Part 3: Between the two double-blind treatment cross-over periods, participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 2) Study Part 4: Participants were crossed-over to second sequence of double-blind treatment (IGIV, 10% or placebo) Study Part 5: Participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 3)
Arm/Group | All Study Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.64 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Grip Strength in the More Affected Hand
Description: The grip strength was measured using a DynEx digital dynamometer. The result of grip strength was recorded to a resolution of 0.1 kg. Each grip strength test consisted of 3 maximal repeated contractions (trials). Each participant will perform 2 sessions of grip strength testing. After a 10-minute break, the testing session will be repeated for a total of 6 grip repetitions per hand.
Time Frame: Week 0, then at Last infusion cycle for each study part (Day 8 of last treatment cycle for 2-week interval or Day 15 of last treatment cycle for 3 or 4 -week interval), then at the end of study visit
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: kilograms
Groups:
- Before Stabilization 1: Baseline Measurements
- End of Stabilization 1: IGIV, 10% (IGIV)
- End of Cross-Over 1: Either IGIV, 10% or Placebo
- End of Stabilization 2; End of Stabilization 3: IGIV, 10%
- End of Cross-Over 2: Either IGIV, 10% or Placebo. The opposite of the end of Cross-Over 1.
- End of the Study: Participants returned following last infusion cycle (2,3, or 4 weeks after last infusion during Stabilization 3) for an End-of-Study visit for assessments including; efficacy (eg: grip strength and disability assessments), adverse events collection, physical examination, laboratory and vital signs, collection and review of diaries and other assessments.
Arm/Group | Before Stabilization 1 | End of Stabilization 1 | End of Cross-Over 1 | End of Stabilization 2 | End of Cross-Over 2 | End of Stabilization 3 | End of the Study
Number analyzed (Participants) | 44 | 44 | 42 | 43 | 43 | 36 | 43
kilograms
  IGIV then Placebo (N= 22, 22, 22, 22, 22, 17, 21) | 18.14 [9.30 to 30.43] | 21.68 [14.05 to 30.83] | 19.54 [10.15 to 29.15] | 19.39 [12.75 to 33.25] | 11.28 [5.50 to 25.92] | 17.77 [9.23 to 27.07] | 17.37 [10.80 to 29.03]
  Placebo then IGIV (N= 22, 22, 20, 21, 21, 19, 22) | 13.17 [5.30 to 20.08] | 14.17 [8.08 to 27.47] | 8.38 [4.86 to 17.03] | 14.18 [7.60 to 27.35] | 15.98 [10.73 to 29.65] | 14.28 [9.47 to 28.25] | 14.00 [7.48 to 24.82]

2. Primary Outcome: Mean Relative Change in Grip Strength in the More Affected Hand
Description: Relative Change is defined as 100 * (End of the Cross-Over Period - baseline of Cross-Over Period) divided by baseline of Cross-Over Period. The grip strength was measured using a DynEx digital dynamometer. The result of grip strength was recorded to a resolution of 0.1 kg. For statistical analysis, the mean of (usually three) trials for cross-over sessions 1 and 2 was computed and the mean of the sessions was used in the analysis as the result of the grip strength measurement. Only if no grip strength testing could be performed the results were considered as missing.
Time Frame: Baseline and last infusion cycle during the two study cross-over periods, approximately weeks 13 and 24; and weeks 37 and 48 (i.e. baseline and end of Study Parts 2 and 4)
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: Percent change in grip strength
Groups:
- Arm 1: IGIV, 10% Then Placebo- Crossover Period 1; Arm 1: IGIV, 10% Then Placebo- Crossover Period 2: Study Part 1: Open-label phase of treatment/stabilization on IGIV, 10% (Stabilization Phase 1) all participants Study Part 2: IGIV, 10% (double-blind treatment cross-over Period 1) Study Part 3: Between the two double-blind treatment cross-over periods, participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 2) Study Part 4: Placebo (0.25% human albumin: BUMINATE 25% Albumin (Human)(Baxter Healthcare Corporation) used where licensed; otherwise Human Albumin 200 g/L Baxter Solution for Infusion was used) (double-blind treatment cross-over Period 2) Study Part 5: Participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 3)
- Arm 2: Placebo Then IGIV, 10% - Crossover Period 1; Arm 2: Placebo Then IGIV, 10% - Crossover Period 2: Study Part 1: Open-label phase of treatment/stabilization on IGIV, 10% (Stabilization Phase 1) all participants Study Part 2: Placebo (0.25% human albumin: BUMINATE 25% Albumin (Human)(Baxter Healthcare Corporation) used where licensed; otherwise Human Albumin 200 g/L Baxter Solution for Infusion was used) (double-blind treatment cross-over Period 1) Study Part 3: Between the two double-blind treatment cross-over periods, participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 2) Study Part 4: IGIV, 10% (double-blind treatment cross-over Period 2) Study Part 5: Participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 3)
Arm/Group | Arm 1: IGIV, 10% Then Placebo- Crossover Period 1 | Arm 1: IGIV, 10% Then Placebo- Crossover Period 2 | Arm 2: Placebo Then IGIV, 10% - Crossover Period 1 | Arm 2: Placebo Then IGIV, 10% - Crossover Period 2
Number analyzed (Participants) | 22 | 22 | 20 | 21
Percent change in grip strength | -16.36 [-30.92 to -1.80] | -30.52 [-43.68 to -17.36] | -30.11 [-48.41 to -11.81] | 23.86 [-23.11 to 70.83]
Statistical Analysis 1: Comparison: Arm 1: IGIV, 10% Then Placebo- Crossover Period 1 vs Arm 1: IGIV, 10% Then Placebo- Crossover Period 2 vs Arm 2: Placebo Then IGIV, 10% - Crossover Period 1 vs Arm 2: Placebo Then IGIV, 10% - Crossover Period 2; Test type: Superiority or Other; p = 0.005, ANOVA; Fixed effects ANOVA with factors for sequence (1 or 2), nested within sequence, period (Cross-Over Period 1 or 2), & treatment (IGIV, 10% or placebo); Difference in least squared means = 35.13, 95% CI 2-sided [8.81 to 61.46]

3. Secondary Outcome: Percentage of Participants With at Least a 30% Decline in Relative Grip Strength in the More Affected Hand (Measured Using a DynEx Digital Dynamometer)
Description: Relative grip strength change is defined as 100 * (End of the Cross-Over Period - baseline of Cross-Over Period) divided by baseline of Cross-Over Period. The grip strength was measured using a DynEx digital dynamometer. The result of grip strength was recorded to a resolution of 0.1 kg. For statistical analysis, the mean of (usually three) trials for cross-over sessions 1 and 2 was computed and the mean of the sessions was used in the analysis as the result of the grip strength measurement. Only if no grip strength testing could be performed the results were considered as missing.
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Number; unit: Percentage of participants
Groups:
- Decline Only During IGIV, 10%: Participants who experienced a relative decrease in grip strength of ≥30% in the more affected hand relative to baseline following IGIV, 10%, but not after the placebo
- Decline Only During Placebo: Participants who experienced a relative decrease in grip strength of ≥30% in the more affected hand relative to baseline following the placebo, but not after IGIV, 10%
- Decline During Both Placebo and IGIV, 10%: Participants who experienced a relative decrease in grip strength of ≥30% in the more affected hand relative to baseline following IGIV, 10%, and the placebo
- No Decline During Placebo or IGIV, 10%: Participants who did not experience a relative decrease in grip strength of ≥30% in the more affected hand relative to baseline following IGIV, 10%, and the placebo
Arm/Group | Decline Only During IGIV, 10% | Decline Only During Placebo | Decline During Both Placebo and IGIV, 10% | No Decline During Placebo or IGIV, 10%
Number analyzed (Participants) | 42 | 42 | 42 | 42
Percentage of participants | 4.8 | 42.9 | 4.8 | 47.6
Statistical Analysis 1: Comparison: Decline Only During IGIV, 10% vs Decline Only During Placebo vs Decline During Both Placebo and IGIV, 10% vs No Decline During Placebo or IGIV, 10%; Test type: Superiority or Other; p < 0.001, McNemar

4. Secondary Outcome: Grip Strength in the Less Affected Hand
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: kilograms
Arm/Group | Before Stabilization 1 | End of Stabilization 1 | End of Cross-Over 1 | End of Stabilization 2 | End of Cross-Over 2 | End of Stabilization 3 | End of the Study
Number analyzed (Participants) | 44 | 44 | 42 | 43 | 43 | 36 | 43
kilograms
  IGIV then Placebo (N= 22, 22, 22, 22, 22, 17, 21) | 27.98 [22.35 to 36.35] | 29.52 [23.28 to 36.98] | 29.79 [20.48 to 37.88] | 29.17 [21.68 to 37.70] | 26.58 [13.67 to 32.83] | 28.97 [15.95 to 34.38] | 29.68 [14.72 to 34.35]
  Placebo then IGIV (N= 22, 22, 20, 21, 21, 19, 22) | 27.23 [18.73 to 34.45] | 28.23 [19.72 to 36.80] | 20.28 [9.61 to 33.44] | 26.92 [17.52 to 37.72] | 27.35 [21.58 to 37.12] | 25.72 [20.18 to 36.55] | 24.98 [16.02 to 35.85]

5. Secondary Outcome: Mean Relative Change in Grip Strength in the Less Affected Hand
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: Percent change in grip strength
Groups:
- Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Cross-over Period 1; Arm 1: IGIV, 10% Then Placebo- Placebo Cross-over Period 2: Study Part 1: Open-label phase of treatment/stabilization on IGIV, 10% (Stabilization Phase 1) all participants Study Part 2: IGIV, 10% (double-blind treatment cross-over Period 1) Study Part 3: Between the two double-blind treatment cross-over periods, participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 2) Study Part 4: Placebo (0.25% human albumin: BUMINATE 25% Albumin (Human)(Baxter Healthcare Corporation) used where licensed; otherwise Human Albumin 200 g/L Baxter Solution for Infusion was used) (double-blind treatment cross-over Period 2) Study Part 5: Participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 3)
- Arm 2: Placebo Then IGIV, 10%- Placebo Cross-over Period 1; Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Cross-over Period 2: Study Part 1: Open-label phase of treatment/stabilization on IGIV, 10% (Stabilization Phase 1) all participants Study Part 2: Placebo (0.25% human albumin: BUMINATE 25% Albumin (Human)(Baxter Healthcare Corporation) used where licensed; otherwise Human Albumin 200 g/L Baxter Solution for Infusion was used) (double-blind treatment cross-over Period 1) Study Part 3: Between the two double-blind treatment cross-over periods, participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 2) Study Part 4: IGIV, 10% (double-blind treatment cross-over Period 2) Study Part 5: Participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 3)
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Cross-over Period 1 | Arm 1: IGIV, 10% Then Placebo- Placebo Cross-over Period 2 | Arm 2: Placebo Then IGIV, 10%- Placebo Cross-over Period 1 | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Cross-over Period 2
Number analyzed (Participants) | 22 | 22 | 20 | 21
Percent change in grip strength | -2.52 [-7.90 to 2.85] | -17.96 [-29.81 to -6.10] | -29.22 [-40.62 to -17.83] | 19.67 [-10.84 to 50.17]
Statistical Analysis 1: Comparison: Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Cross-over Period 1 vs Arm 1: IGIV, 10% Then Placebo- Placebo Cross-over Period 2 vs Arm 2: Placebo Then IGIV, 10%- Placebo Cross-over Period 1 vs Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Cross-over Period 2; Test type: Superiority or Other; p < 0.001, ANOVA; Difference in least squared means = 32.54, 95% CI 2-sided [14.01 to 51.06]

6. Secondary Outcome: Proportion of Participants That Were Accelerated Forward Into the Next Stabilization Phase (ie Switched to Open-Label IGIV, 10%)
Description: Participants were permitted to switch from blinded treatment with placebo or IGIV, 10% to open label IGIV, 10% if they and investigator agreed that deterioration had occurred to the extent that the participant had unacceptable difficulty carrying out daily activities involving the affected muscles, or decline in grip strength of ≥50% in the more affected hand had occurred.
Time Frame: During the two study cross-over periods, approximately weeks 13-24 and weeks 37-48 (i.e. Study Parts 2 and 4)
Population: Intent to treat
Measure: Number; unit: Proportion of participants
Groups:
- Accelerated Switch During IGIV, 10% and Placebo: Participants who required a switch to open label IGIV, 10% when receiving IGIV, 10%, and placebo
- Accelerated Switch During Placebo, But Not IGIV, 10%: Participants who required a switch to open label IGIV, 10% when receiving the placebo, but not during IGIV, 10%
- Accelerated Switch During IGIV, 10%, But Not Placebo: Participants who required a switch to open label IGIV, 10% when receiving IGIV, 10%, but not during placebo
- No Accelerated Switch During IGIV, 10% or Placebo: Participants who did not require a switch to open label IGIV, 10% when receiving IGIV, 10%, or placebo
Arm/Group | Accelerated Switch During IGIV, 10% and Placebo | Accelerated Switch During Placebo, But Not IGIV, 10% | Accelerated Switch During IGIV, 10%, But Not Placebo | No Accelerated Switch During IGIV, 10% or Placebo
Number analyzed (Participants) | 42 | 42 | 42 | 42
Proportion of participants | 0.0 | 69.0 | 2.4 | 28.6
Statistical Analysis 1: Comparison: Accelerated Switch During IGIV, 10% and Placebo vs Accelerated Switch During Placebo, But Not IGIV, 10% vs Accelerated Switch During IGIV, 10%, But Not Placebo vs No Accelerated Switch During IGIV, 10% or Placebo; Test type: Superiority or Other; p < 0.001, McNemar

7. Secondary Outcome: Patient Global Impression of Change
Description: Patient Global Impression of Change was measured on an ordinal scale of 1-7, higher scores representing greater perceived deterioration since the previous efficacy assessment (ranging from (1) very much improved to very much worse (7)). 1. Very much improved 2. Much improved 3. Minimally improved 4. No change 5. Minimally worse 6. Much worse 7. Very much worse
Time Frame: Last infusion cycle for each study part (Day 8 of last treatment cycle for 2-week interval or Day 15 of last treatment cycle for 3 or 4 -week interval), then at the end of study visit
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Groups:
- End of Stabilization 1; End of Stabilization 2; End of Stabilization 3: (IGIV, 10%)
Arm/Group | End of Stabilization 1 | End of Cross-Over 1 | End of Stabilization 2 | End of Cross-Over 2 | End of Stabilization 3 | End of the Study
Number analyzed (Participants) | 44 | 42 | 43 | 43 | 36 | 43
Scores on a scale
  IGIV, 10% then Placebo (N= 22, 22, 22, 21, 17, 21) | 4.0 [3.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 5.0 [5.0 to 6.0] | 2.0 [2.0 to 4.0] | 4.0 [3.0 to 4.0]
  Placebo then IGIV, 10% (N= 22, 20, 21, 21, 19, 22) | 4.0 [3.0 to 4.0] | 6.0 [5.0 to 6.0] | 3.0 [2.0 to 3.0] | 4.0 [3.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]

8. Secondary Outcome: Overall Disability Sum Score
Description: The overall disability sum scale (based on Merkies et al., 2002) is a patient questionnaire that measures disability. Overall disability sum score = arm disability scale (range 0-5) + leg disability scale (range 0-7); Overall Range: 0 (no signs of disability) to 12 (maximum disability).
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Before Stabilization 1 | End of Stabilization 1 | End of Cross-Over 1 | End of Stabilization 2 | End of Cross-Over 2 | End of Stabilization 3 | End of the Study
Number analyzed (Participants) | 44 | 44 | 42 | 43 | 43 | 36 | 43
Scores on a scale
  IGIV then Placebo (N= 22, 22, 22, 22, 22, 17, 21) | 3 [2 to 4] | 2 [2 to 4] | 3 [2 to 4] | 2 [2 to 4] | 3 [2 to 4] | 2 [2 to 4] | 2 [2 to 4]
  Placebo then IGIV (N= 22, 22, 20, 21, 21, 19, 22) | 3 [2 to 4] | 3 [2 to 4] | 4 [3 to 5] | 3 [2 to 4] | 3 [2 to 4] | 4 [2 to 4] | 3 [2 to 4]

9. Secondary Outcome: Overall Disability Sum Score - Standardized
Description: The overall disability sum scale (based on Merkies et al., 2002) is a patient questionnaire that measures disability. Overall disability sum score = arm disability scale (range 0-5) + leg disability scale (range 0-7); Overall Range: 0 (no signs of disability) to 12 (maximum disability). This was standardized to a scale of 0 to 100 (the best score being 100) to allow calculation of relative changes.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Before Stabilization 1 | End of Stabilization 1 | End of Cross-Over 1 | End of Stabilization 2 | End of Cross-Over 2 | End of Stabilization 3 | End of the Study
Number analyzed (Participants) | 44 | 44 | 42 | 43 | 43 | 36 | 43
Scores on a scale
  IGIV then Placebo (N= 22, 22, 22, 22, 22, 17, 21) | 75.0 [66.7 to 83.3] | 83.3 [66.7 to 83.3] | 79.2 [66.7 to 83.3] | 83.3 [66.7 to 83.3] | 75.0 [66.7 to 83.3] | 83.3 [66.7 to 83.3] | 83.3 [66.7 to 83.3]
  Placebo then IGIV (N= 22, 22, 20, 21, 21, 19, 22) | 75.0 [66.7 to 83.3] | 75.0 [66.7 to 83.3] | 66.7 [58.3 to 75.0] | 75.0 [66.7 to 83.3] | 75.0 [66.7 to 83.3] | 66.7 [66.7 to 83.3] | 75.0 [66.7 to 83.3]

10. Secondary Outcome: Mean Relative Change in Overall Disability Sum Score
Description: Relative Change is defined as 100 * (End of the Cross-Over Period - baseline of Cross-Over Period) divided by baseline of Cross-Over Period. The overall disability sum scale (based on Merkies et al., 2002) is a patient questionnaire that measures disability (from 0, "no signs of disability" to 12, "most severe disability"). This was standardized to a scale of 0 to 100 (the best score being 100) to allow calculation of relative changes.
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: percent change in score
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Cross-over Period 1 | Arm 1: IGIV, 10% Then Placebo- Placebo Cross-over Period 2 | Arm 2: Placebo Then IGIV, 10%- Placebo Cross-over Period 1 | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Cross-over Period 2
Number analyzed (Participants) | 22 | 22 | 20 | 21
percent change in score | -3.14 [-6.55 to 0.27] | -5.77 [-10.33 to -1.20] | -8.46 [-12.81 to -4.11] | 0.92 [-2.88 to 4.73]
Statistical Analysis 1: Comparison: Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Cross-over Period 1 vs Arm 1: IGIV, 10% Then Placebo- Placebo Cross-over Period 2 vs Arm 2: Placebo Then IGIV, 10%- Placebo Cross-over Period 1 vs Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Cross-over Period 2; Test type: Superiority or Other; p = 0.002, ANOVA; Difference in Least Squared Means = 6.03, 95% CI 2-sided [2.14 to 9.92]

11. Secondary Outcome: Time Required by Participants to Complete the 9 Hole Peg Board Test (9-HPT) With the Dominant Hand
Description: The 9-HPT is a quantitative measure of upper extremity (arm and hand) function. Participants picked up the pegs one at a time (nine in total), and put them into the holes on the board as quickly as possible, in any order until all the holes were filled. Then, without pausing, participants removed the pegs one at a time and returned them to the container as quickly as possible. Each participant did this two times with their dominant hand. The 9-HCT objective is to see how fast participants could put all of the pegs in and take them out again.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Before Stabilization 1 | End of Stabilization 1 | End of Cross-Over 1 | End of Stabilization 2 | End of Cross-Over 2 | End of Stabilization 3 | End of the Study
Number analyzed (Participants) | 44 | 44 | 42 | 43 | 43 | 36 | 43
Seconds
  IGIV then Placebo (N= 22, 22, 22, 22, 22, 17, 21) | 20.75 [19.50 to 27.50] | 22.00 [19.50 to 29.00] | 20.25 [18.00 to 29.00] | 21.00 [18.00 to 24.50] | 20.50 [18.50 to 27.50] | 20.50 [19.00 to 24.50] | 20.00 [19.00 to 25.50]
  Placebo then IGIV (N= 22, 22, 20, 21, 21, 19, 22) | 26.75 [20.50 to 39.00] | 25.25 [19.00 to 33.50] | 27.75 [23.00 to 43.50] | 24.50 [19.00 to 34.50] | 25.00 [20.00 to 30.50] | 27.50 [20.50 to 35.50] | 26.25 [19.50 to 33.00]

12. Secondary Outcome: Mean Relative Change in Time Required by Participants to Complete the 9 Hole Peg Board Test (9-HPT) With the Dominant Hand
Description: Relative Change is defined as 100 * (End of the Cross-Over Period - baseline of Cross-Over Period) divided by baseline of Cross-Over Period. The 9-HPT is a quantitative measure of upper extremity (arm and hand) function. Participants picked up the pegs one at a time (nine in total), and put them into the holes on the board as quickly as possible, in any order until all the holes were filled. Then, without pausing, participants removed the pegs one at a time and returned them to the container as quickly as possible. Each participant did this two times with their dominant hand. The 9-HCT objective is to see how fast participants could put all of the pegs in and take them out again.
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: Percent change in time
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Cross-over Period 1 | Arm 1: IGIV, 10% Then Placebo- Placebo Cross-over Period 2 | Arm 2: Placebo Then IGIV, 10%- Placebo Cross-over Period 1 | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Cross-over Period 2
Number analyzed (Participants) | 22 | 22 | 20 | 21
Percent change in time | -2.57 [-9.99 to 4.86] | 3.90 [-4.59 to 12.39] | 29.89 [12.46 to 47.31] | 4.89 [-9.45 to 19.23]
Statistical Analysis 1: Comparison: Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Cross-over Period 1 vs Arm 1: IGIV, 10% Then Placebo- Placebo Cross-over Period 2 vs Arm 2: Placebo Then IGIV, 10%- Placebo Cross-over Period 1 vs Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Cross-over Period 2; Test type: Superiority or Other; p < 0.001, ANOVA; Difference in Least Squared Means = -15.57, 95% CI 2-sided [-24.37 to -6.77]

13. Secondary Outcome: Time Required by Participants to Complete the 9 Hole Peg Board Test (9-HPT) With the Non-Dominant Hand
Description: The 9-HPT is a quantitative measure of upper extremity (arm and hand) function. Participants picked up the pegs one at a time (nine in total), and put them into the holes on the board as quickly as possible, in any order until all the holes were filled. Then, without pausing, participants removed the pegs one at a time and returned them to the container as quickly as possible. Each participant did this two times with their non-dominant hand. The 9-HCT objective is to see how fast participants could put all of the pegs in and take them out again.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Before Stabilization 1 | End of Stabilization 1 | End of Cross-Over 1 | End of Stabilization 2 | End of Cross-Over 2 | End of Stabilization 3 | End of the Study
Number analyzed (Participants) | 44 | 44 | 42 | 43 | 43 | 36 | 43
Seconds
  IGIV then Placebo (N= 22, 22, 22, 22, 22, 17, 21) | 25.75 [20.00 to 29.50] | 22.50 [19.50 to 27.00] | 24.00 [19.50 to 28.50] | 23.50 [19.50 to 27.00] | 25.25 [22.50 to 29.50] | 21.00 [19.50 to 24.50] | 23.00 [20.50 to 26.50]
  Placebo then IGIV (N= 22, 22, 20, 21, 21, 19, 22) | 31.25 [22.50 to 51.00] | 28.00 [22.50 to 40.00] | 37.25 [26.25 to 82.75] | 31.50 [24.00 to 38.50] | 32.50 [22.00 to 41.00] | 30.00 [22.50 to 39.50] | 30.00 [21.00 to 38.50]

14. Secondary Outcome: Mean Relative Change in Time Required by Participants to Complete the 9 Hole Peg Board Test (9-HPT) With the Non-Dominant Hand
Description: Relative Change is defined as 100 * (End of the Cross-Over Period - baseline of Cross-Over Period) divided by baseline of Cross-Over Period. The 9-HPT is a quantitative measure of upper extremity (arm and hand) function. Participants picked up the pegs one at a time (nine in total), and put them into the holes on the board as quickly as possible, in any order until all the holes were filled. Then, without pausing, participants removed the pegs one at a time and returned them to the container as quickly as possible. Each participant did this two times with their non-dominant hand. The 9-HCT objective is to see how fast participants could put all of the pegs in and take them out again.
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: Percent change in time
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Cross-over Period 1 | Arm 1: IGIV, 10% Then Placebo- Placebo Cross-over Period 2 | Arm 2: Placebo Then IGIV, 10%- Placebo Cross-over Period 1 | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Cross-over Period 2
Number analyzed (Participants) | 22 | 22 | 20 | 21
Percent change in time | 4.78 [-1.65 to 11.21] | 13.06 [4.46 to 21.65] | 52.93 [26.82 to 79.05] | 8.56 [-4.88 to 22.01]
Statistical Analysis 1: Comparison: Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Cross-over Period 1 vs Arm 1: IGIV, 10% Then Placebo- Placebo Cross-over Period 2 vs Arm 2: Placebo Then IGIV, 10%- Placebo Cross-over Period 1 vs Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Cross-over Period 2; Test type: Superiority or Other; p < 0.001, ANOVA; Difference in Least Squared Means = -26.11, 95% CI 2-sided [-38.96 to -13.26]

15. Secondary Outcome: Participants' Assessment of Physical Functioning on a Visual Analog Scale (VAS)
Description: The VAS measured patients' assessment of physical functioning on a 10 centimeter scale of 0-10, on which 0 represents "no symptoms" and 10 "disabled, unable to use affected limbs".
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Before Stabilization 1 | End of Stabilization 1 | End of Cross-Over 1 | End of Stabilization 2 | End of Cross-Over 2 | End of Stabilization 3 | End of the Study
Number analyzed (Participants) | 44 | 44 | 42 | 43 | 43 | 36 | 43
Scores on a scale
  IGIV then Placebo (N= 22, 22, 22, 22, 22, 17, 21) | 4.80 [2.90 to 6.30] | 2.95 [1.60 to 5.10] | 4.10 [2.00 to 5.60] | 3.50 [1.70 to 5.10] | 6.85 [5.90 to 8.10] | 4.50 [2.60 to 5.10] | 3.70 [1.90 to 5.40]
  Placebo then IGIV (N= 22, 22, 20, 21, 21, 19, 22) | 4.95 [2.30 to 7.60] | 3.15 [2.70 to 5.50] | 7.15 [6.75 to 7.60] | 5.10 [2.30 to 6.10] | 4.60 [2.40 to 5.90] | 4.50 [2.60 to 6.00] | 5.15 [2.80 to 6.30]

16. Secondary Outcome: Mean Relative Change in Participants' Assessment of Physical Functioning on a Visual Analog Scale (VAS)
Description: Relative Change is defined as 100 * (End of the Cross-Over Period - baseline of Cross-Over Period) divided by baseline of Cross-Over Period. The VAS measured patients' assessment of physical functioning on a 10 centimeter scale of 0-10, on which 0 represents "no symptoms" and 10 "disabled, unable to use affected limbs".
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: Percent change in assessment
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Cross-over Period 1 | Arm 1: IGIV, 10% Then Placebo- Placebo Cross-over Period 2 | Arm 2: Placebo Then IGIV, 10%- Placebo Cross-over Period 1 | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Cross-over Period 2
Number analyzed (Participants) | 22 | 22 | 20 | 21
Percent change in assessment | 140.92 [-1.35 to 283.19] | 321.75 [-73.45 to 716.95] | 258.09 [-100.83 to 617.01] | 5.75 [-11.54 to 23.04]
Statistical Analysis 1: Comparison: Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Cross-over Period 1 vs Arm 1: IGIV, 10% Then Placebo- Placebo Cross-over Period 2 vs Arm 2: Placebo Then IGIV, 10%- Placebo Cross-over Period 1 vs Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Cross-over Period 2; Test type: Superiority or Other; p = 0.059, ANOVA; Difference in Least Squared Means = -216.60, 95% CI 2-sided [-490.41 to 57.22]

17. Primary Outcome: Co-Primary Endpoint: Guy's Neurologic Disability Scale (GNDS) for Upper Limbs
Description: GNDS (based on Sharrack and Hughes, 1999) for the upper limbs were integers 0 to 5, with 0 indicating no impairment.
Time Frame: as for outcome 1
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Before Stabilization 1 | End of Stabilization 1 | End of Cross-Over 1 | End of Stabilization 2 | End of Cross-Over 2 | End of Stabilization 3 | End of the Study
Number analyzed (Participants) | 44 | 44 | 42 | 43 | 43 | 36 | 43
Scores on a scale
  IGIV then Placebo (N= 22, 22, 22, 22, 22, 17, 21) | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 3.0] | 2.5 [2.0 to 3.0] | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 2.0]
  Placebo then IGIV (N= 22, 22, 20, 21, 21, 19, 22) | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]

18. Post Hoc Outcome: Proportion of Participants With at Least a 30% Decline in Relative Grip Strength in the Less Affected Hand (Measured Using a DynEx Digital Dynamometer)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Number; unit: Proportion of participants
Groups:
- Decline Only During IGIV, 10%: Participants who experienced a relative decrease in grip strength of ≥30% in the less affected hand relative to baseline following IGIV, 10%, but not after the placebo
- Decline Only During Placebo: Participants who experienced a relative decrease in grip strength of ≥30% in the less affected hand relative to baseline following the placebo, but not after IGIV, 10%
- Decline During Both Placebo and IGIV, 10%: Participants who experienced a relative decrease in grip strength of ≥30% in the less affected hand relative to baseline following IGIV, 10%, and the placebo
- No Decline During Placebo and IGIV, 10%: Participants who did not experience a relative decrease in grip strength of ≥30% in the less affected hand relative to baseline following IGIV, 10%, and the placebo
Arm/Group | Decline Only During IGIV, 10% | Decline Only During Placebo | Decline During Both Placebo and IGIV, 10% | No Decline During Placebo and IGIV, 10%
Number analyzed (Participants) | 42 | 42 | 42 | 42
Proportion of participants | 0.0 | 31.0 | 2.4 | 66.7
Statistical Analysis 1: Comparison: Decline Only During IGIV, 10% vs Decline Only During Placebo vs Decline During Both Placebo and IGIV, 10% vs No Decline During Placebo and IGIV, 10%; Test type: Superiority or Other; p < 0.001, McNemar

19. Primary Outcome: Co-Primary Endpoint: Proportion of Participants With Deterioration in Guy's Neurological Disability Score (GNDS)
Description: GNDS (based on Sharrack and Hughes, 1999) for the upper limbs were integers 0 to 5, with 0 indicating no impairment.
Time Frame: as for outcome 2
Population: Intent to treat
Measure: Number; unit: Proportion of participants
Groups:
- Deterioration After IGIV, 10% and Placebo: Participants with deterioration in GNDS scores after IGIV, 10% and placebo
- Deterioration After Placebo, But Not IGIV, 10%: Participants with deterioration in GNDS scores after Placebo, but not IGIV, 10%
- Deterioration After IGIV, 10%, But Not Placebo: Participants with deterioration in GNDS scores after IGIV, 10%, but not Placebo
- No Deterioration After IGIV, 10% or Placebo: Participants with no deterioration in GNDS scores after IGIV, 10% or Placebo
Arm/Group | Deterioration After IGIV, 10% and Placebo | Deterioration After Placebo, But Not IGIV, 10% | Deterioration After IGIV, 10%, But Not Placebo | No Deterioration After IGIV, 10% or Placebo
Number analyzed (Participants) | 42 | 42 | 42 | 42
Proportion of participants | 4.8 [2.0 to 2.0] | 35.7 [2.0 to 3.0] | 11.9 [2.0 to 3.0] | 47.6 [2.0 to 3.0]
Statistical Analysis 1: Comparison: Deterioration After IGIV, 10% and Placebo vs Deterioration After Placebo, But Not IGIV, 10% vs Deterioration After IGIV, 10%, But Not Placebo vs No Deterioration After IGIV, 10% or Placebo; Test type: Superiority or Other; p = 0.021, McNemar

20. Primary Outcome: Rate of Temporally Associated Adverse Events (AEs) Per Infusion
Description: The total number of all AEs which begin during or within 72 hours of completion of an infusion, irrespective of being related or not related to the study product (IGIV, 10% or Placebo), divided by the total number of infusions, and multiplied by 100.
Time Frame: Within 72 hours of completion of an infusion during the two study cross-over periods, approximately weeks 13-24 and weeks 37-48 (i.e. Study Parts 2 and 4)
Population: Safety Dataset
Measure: Number; unit: Percentage of AEs per infusion
Units Other Than Participants: Infusions
Groups:
- Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Period; Arm 1: IGIV, 10% Then Placebo- Placebo Period: Study Part 1: Open-label phase of treatment/stabilization on IGIV, 10% (Stabilization Phase 1) all participants Study Part 2: IGIV, 10% (double-blind treatment cross-over Period 1) Study Part 3: Between the two double-blind treatment cross-over periods, participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 2) Study Part 4: Placebo (0.25% human albumin: BUMINATE 25% Albumin (Human)(Baxter Healthcare Corporation) used where licensed; otherwise Human Albumin 200 g/L Baxter Solution for Infusion was used) (double-blind treatment cross-over Period 2) Study Part 5: Participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 3)
- Arm 2: Placebo Then IGIV, 10%- Placebo Period; Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Period: Study Part 1: Open-label phase of treatment/stabilization on IGIV, 10% (Stabilization Phase 1) all participants Study Part 2: Placebo (0.25% human albumin: BUMINATE 25% Albumin (Human)(Baxter Healthcare Corporation) used where licensed; otherwise Human Albumin 200 g/L Baxter Solution for Infusion was used) (double-blind treatment cross-over Period 1) Study Part 3: Between the two double-blind treatment cross-over periods, participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 2) Study Part 4: IGIV, 10% (double-blind treatment cross-over Period 2) Study Part 5: Participants received open-label treatment/stabilization with IGIV, 10% for 12 weeks (Stabilization Phase 3)
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Period | Arm 1: IGIV, 10% Then Placebo- Placebo Period | Arm 2: Placebo Then IGIV, 10%- Placebo Period | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Period
Number analyzed (Participants) | 22 | 22 | 21 | 21
Number analyzed (Infusions) | 104 | 68 | 61 | 138
Percentage of AEs per infusion | 11.5 | 13.2 | 24.6 | 11.6

21. Primary Outcome: The Percentage of Participants for Whom the Infusion Rate of Any Infusion Was Reduced and/or the Infusion Was Interrupted or Stopped for Any Reason
Time Frame: Throughout the two study cross-over periods, approximately weeks 13-24 and weeks 37-48 (i.e. Study Parts 2 and 4)
Population: Safety Dataset
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Period | Arm 1: IGIV, 10% Then Placebo- Placebo Period | Arm 2: Placebo Then IGIV, 10%- Placebo Period | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Period
Number analyzed (Participants) | 22 | 22 | 21 | 21
percentage of participants | 9.1 | 0.0 | 4.8 | 4.8

22. Primary Outcome: The Percentage of Infusions for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped for Any Reason
Time Frame: Throughout the two study cross-over periods, approximately weeks 13-24 and weeks 37-48 (i.e. Study Parts 2 and 4)
Population: Safety Dataset
Measure: Number; unit: percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Period | Arm 1: IGIV, 10% Then Placebo- Placebo Period | Arm 2: Placebo Then IGIV, 10%- Placebo Period | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Period
Number analyzed (Participants) | 22 | 22 | 21 | 21
Number analyzed (Infusions) | 104 | 68 | 61 | 138
percentage of infusions | 2.9 | 0.0 | 1.6 | 0.7

23. Secondary Outcome: Rate of Related AEs Per Infusion
Description: The total number of AEs determined by the investigator to be related to the study product that occur at any time during the study divided by the total number of infusions, and multiplied by 100.
Time Frame: Throughout the two study cross-over periods, approximately weeks 13-24 and weeks 37-48 (i.e. Study Parts 2 and 4)
Population: Safety Dataset
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Period | Arm 1: IGIV, 10% Then Placebo- Placebo Period | Arm 2: Placebo Then IGIV, 10%- Placebo Period | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Period
Number analyzed (Participants) | 22 | 22 | 21 | 21
Number analyzed (Infusions) | 104 | 68 | 61 | 138
AEs per infusion | 4.8 | 20.6 | 44.3 | 15.9

24. Secondary Outcome: Rate of Related SAEs Per Infusion
Description: The total number of SAEs determined by the investigator to be related to the study product that occur at any time during the study divided by the total number of infusions, and multiplied by 100.
Time Frame: Throughout the two study cross-over periods, approximately weeks 13-24 and weeks 37-48 (i.e. Study Parts 2 and 4)
Population: Safety Dataset
Measure: Number; unit: SAEs per infusion
Units Other Than Participants: Infusions
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Period | Arm 1: IGIV, 10% Then Placebo- Placebo Period | Arm 2: Placebo Then IGIV, 10%- Placebo Period | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Period
Number analyzed (Participants) | 22 | 22 | 21 | 21
Number analyzed (Infusions) | 104 | 68 | 61 | 138
SAEs per infusion | 0.0 | 0.0 | 0.0 | 0.7

25. Secondary Outcome: The Proportion of Participants for Whom the Infusion Rate of Any Infusion Was Reduced and/or the Infusion Was Interrupted or Stopped for Tolerability Concerns/AEs
Time Frame: Throughout the two study cross-over periods, approximately weeks 13-24 and weeks 37-48 (i.e. Study Parts 2 and 4)
Population: Safety Dataset
Measure: Number; unit: proportion of participants
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Period | Arm 1: IGIV, 10% Then Placebo- Placebo Period | Arm 2: Placebo Then IGIV, 10%- Placebo Period | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Period
Number analyzed (Participants) | 22 | 22 | 21 | 21
proportion of participants | 0.0 | 0.0 | 0.0 | 4.8

26. Secondary Outcome: The Proportion of Infusions for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped for Tolerability Concerns/AEs
Time Frame: Throughout the two study cross-over periods, approximately weeks 13-24 and weeks 37-48 (i.e. Study Parts 2 and 4)
Population: Safety Dataset
Measure: Number; unit: proportion of infusions
Units Other Than Participants: Infusions
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Period | Arm 1: IGIV, 10% Then Placebo- Placebo Period | Arm 2: Placebo Then IGIV, 10%- Placebo Period | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Period
Number analyzed (Participants) | 22 | 22 | 21 | 21
Number analyzed (Infusions) | 104 | 68 | 61 | 138
proportion of infusions | 0.0 | 0.0 | 0.0 | 0.7

27. Secondary Outcome: The Proportion of Infusions Associated With One or More AEs Related to the Study Product
Time Frame: Throughout the two study cross-over periods, approximately weeks 13-24 and weeks 37-48 (i.e. Study Parts 2 and 4)
Population: Safety Dataset
Measure: Number; unit: proportion of infusions
Units Other Than Participants: Infusions
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Period | Arm 1: IGIV, 10% Then Placebo- Placebo Period | Arm 2: Placebo Then IGIV, 10%- Placebo Period | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Period
Number analyzed (Participants) | 22 | 22 | 21 | 21
Number analyzed (Infusions) | 104 | 68 | 61 | 138
proportion of infusions | 3.8 | 19.1 | 34.4 | 13.0

28. Primary Outcome: The Percentage of Participants Reporting One or More Moderate or Severe AEs That Began During Infusion or Within 72 Hours of Completion of an Infusion
Time Frame: as for outcome 20
Population: Safety Dataset
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: IGIV, 10% Then Placebo- IGIV, 10% Period | Arm 1: IGIV, 10% Then Placebo- Placebo Period | Arm 2: Placebo Then IGIV, 10%- Placebo Period | Arm 2: Placebo Then IGIV, 10%- IGIV, 10% Period
Number analyzed (Participants) | 22 | 22 | 21 | 21
percentage of participants | 4.5 | 27.3 | 19.0 | 4.8

ADVERSE EVENTS:
Time Frame: Throughout the study period, approximately three years.
Groups:
- IGIV, 10%: Participants received IGIV, 10% at the same equivalent dose per week administered prior to the study (0.4 to 2.0 g per kg BW per infusion cycle)
- Placebo: 0.25% human albumin: BUMINATE 25% Albumin (Human)(Baxter Healthcare Corporation) used where licensed; otherwise Human Albumin 200 g/L Baxter Solution for Infusion was used)
Arm/Group | IGIV, 10% | Placebo
Serious Adverse Events (participants affected / at risk) | 2/44 | 0/43
Other Adverse Events (participants affected / at risk) | 35/44 | 33/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV, 10% (N=44) | Placebo (N=43)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV, 10% (N=44) | Placebo (N=43)
HEADACHE (Nervous system disorders) | 16 (34) | 2 (3)
NEUROLOGICAL DECOMPENSATION (Nervous system disorders) | 10 (10) | 25 (25)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (15) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 8 (12) | 2 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 7 (9) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 6 (9) | 2 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (2)
CONTUSION (Injury, poisoning and procedural complications) | 5 (9) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (6) | 3 (3)
CHEST DISCOMFORT (General disorders) | 3 (3) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 0 (0)
FATIGUE (General disorders) | 3 (5) | 0 (0)
NASOPHARYNGITIS (General disorders) | 3 (3) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 3 (31) | 2 (3)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 3 (3) | 2 (2)
PARAESTHESIA (Nervous system disorders) | 3 (4) | 1 (1)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
SINUS HEADACHE (Nervous system disorders) | 3 (3) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 3 (3) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 18 months after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥90 days prior to submission or communication. Baxter may request an additional delay of ≤120 days(e.g., for intellectual property protection)